CLINICAL TRIAL: NCT04718207
Title: Interest of PFS Modelling in the Quantitative Analysis of Brain PET Scans in Patients With Alzheimer's Disease Acquired on a Numerical System
Brief Title: Modelling in the Quantitative Analysis of Brain PET Scans in Patients With Alzheimer's Disease
Acronym: PET-SF
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, PU-PH, Central Hospital, Nancy, France
Other Study IDs: S201215_051
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Patients With Alzheimer's Disease
Keywords: Alzheimer disease; PSF modelisation; quantitative analyze
MeSH Terms: conditions — Alzheimer Disease | interventions — Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Alzheimer disease: Patients recruited retrospectively with the available nuclear medicine listing of patients who performed brain PET/CT scans in the nuclear medicine department from December 2017 to December 2020.
  Interventions: Device: Brain positron emission tomopgraphy (PET) - scan

INTERVENTIONS:
Device: Brain positron emission tomopgraphy (PET) - scan — Patients who performed brain PET/CT scans in the nuclear medicine department from December 2017 to December 2020.

SUMMARY:
PET/CT scans with 18F-FDG can be carried out for the detection of neurodegenerative diseases with hypometabolisms characteristic of the pathologies sought. The diagnosis is given by the clinician after a visual analysis of the data. To complete the diagnosis, a semi-quantitative analysis of the images is recommended (European recommendations) in addition to the visual analysis.

DETAILED DESCRIPTION:
PET/CT scans with 18F-FDG can be carried out for the detection of neurodegenerative diseases with hypometabolisms characteristic of the pathologies sought. The diagnosis is given by the clinician after a visual analysis of the data. To complete the diagnosis, a semi-quantitative analysis of the images is recommended (European recommendations) in addition to the visual analysis.

PET technology is improving from year to year thanks to the arrival of a new PET technology called digital. In addition, correction methods have been developed to improve PET images and thus improve the detection of different pathologies in PET.

The PSF (Point Spread Function) tool enables partial volume effects to be corrected. The PSF consists of correcting the impulse response of the system, and allows a visual improvement of the images. Currently not recommended in brain PET/CT reconstructions, it remains to be evaluated for the quantitative analysis of acquisitions.

ELIGIBILITY:
Inclusion Criteria:

* Brain PET/CT scans at 18F-FDG of patients with Alzheimer's disease carried out in the nuclear medicine department of the Nancy-Brabois University Hospital since December 2017 on digital PET devices.

Exclusion Criteria:

* Patients who have expressed their opposition to the use of their data (poster in the service).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Alzheimer disease
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
The results obtained in quantitative analysis with and without PSF modelling of PET brain scans of patients with Alzheimer's disease acquired on PET / CT scan | 6 months
  Comparison of the volumes detected by the quantitative analysis with the SPM (statistical parametric Mapping) software of brain PET scans of patients with Alzheimer's disease with and without FSP modelling.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuclear medicine department CHRU de NANCY Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No